CLINICAL TRIAL: NCT06086795
Title: Investigating Age-dependent Effects of Egg Intake on HDL and Immune Profiles
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Catherine Andersen, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H22-0174; AG221113 (Other Grant/Funding Number: American Egg Board)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Lipoproteins; Inflammatory Response
Keywords: Diet; Lipoproteins; T-Lymphocytes; Eggs; Aging
MeSH Terms: interventions — Egg Yolk; Egg White

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Egg whites (Active Comparator): 3 large egg equivalent of liquid egg whites per day for 4 weeks
  Interventions: Other: Egg whites
- Egg yolks (Experimental): 3 large egg equivalent of liquid egg yolks per day for 4 weeks
  Interventions: Other: Egg yolks
- Whole eggs (Experimental): 3 large whole eggs per day for 4 weeks
  Interventions: Other: Whole eggs

INTERVENTIONS:
Other: Whole eggs — 3 large whole eggs per day for 4 weeks
  Arms: Whole eggs
Other: Egg yolks — 3 large egg equivalent of egg yolks per day for 4 weeks
  Arms: Egg yolks
Other: Egg whites — 3 large egg equivalent of egg whites per day for 4 weeks
  Arms: Egg whites

SUMMARY:
The goal of this intervention study is to determine whether consumption of different fractions of chicken eggs, including egg whites, egg yolks, and whole eggs, confer different changes in markers of HDL function and T cell profiles in younger vs. older men and women. The study will address the following objectives:

* Objective 1: Determine if daily consumption of egg fractions differentially alter HDL profiles across age groups.
* Objective 2: Determine if daily consumption of egg fractions differentially alter immune cell profiles across age groups.

Participants will be asked to consume egg whites, egg yolks, and whole eggs on a daily basis for 4-weeks each, and avoid eating eggs for a total of 8 weeks at different points in the study. Participants will additionally be provided guidance on following a generally healthy diet, and will be asked to complete surveys about dietary intake and physical activity, as well as provide blood samples throughout the course of the study.

Researchers will compare whether daily consumption of egg whites, egg yolks, and whole eggs differentially alter markers of HDL function and T cell profiles in younger vs. older adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old, or 50-75 years old (at time of screening)
* Body mass index (BMI) < 30 kg/m2
* Willing to consume whole eggs, egg whites, or egg yolks on a daily basis during study periods, and refrain from eating eggs during other study periods
* Do not fit any exclusion criteria

Exclusion Criteria:

* < 18 years old; 31-49 years old; > 75 years old
* BMI ≥ 30 kg/m2 or body weight < 110 pounds
* Weight changes > 10% over the last 4 weeks
* Self-reported history of diabetes, heart disease, stroke, renal or liver disease, cancer, eating disorders, certain severe and/or relapsing/remitting autoimmune, inflammatory, or metabolic diseases, chronic infections, scleroderma, blood clotting disorders, intravenous drug use, or current pregnancy or lactation
* Allergy or intolerance to eggs, egg components, or egg products
* Implanted medical device (e.g., pacemaker) or other health condition that would prevent measurement of body composition by bioelectrical impedance
* Highly elevated fasting lipid and glucose levels (triglyceride levels higher than 500 mg/dL, fasting glucose higher than 126 mg/dL), or total cholesterol < 120 mg/dL and HDL-cholesterol < 15 mg/dL
* Currently taking lipid-lowering medications (e.g. statins, fibrates), anti-inflammatory medications (e.g., NSAIDs, corticosteroids), or medications that primarily affect blood clotting (e.g., warfarin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum concentration of large HDL particles between diet periods | 4 weeks
  Measurement of serum large HDL particles (nmol/L) at the egg-free run-in period and the end of each intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Andersen, PhD, RDN, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No